CLINICAL TRIAL: NCT02608710
Title: A Phase 1, Randomized, Open-Label Study in Healthy Adult Male Subjects to Assess the Pharmacokinetics and Pharmacodynamics of RDEA3170
Brief Title: RDEA3170 PK/PD Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA3170-112
Record Dates: First submitted 2015-11-15; First posted 2015-11-20 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — verinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single Dose (Experimental): Single dose of RDEA3170 4.5 mg, RDEA3170 6 mg or RDEA3170 12 mg on Days 1, 5 and 9.
  Interventions: Drug: RDEA3170 4.5 mg; Drug: RDEA3170 6 mg; Drug: RDEA3170 12 mg
- Multiple Dose (Experimental): RDEA3170 12 mg once daily (qd)
  Interventions: Drug: RDEA3170 12 mg
- Single Dose Food Effect (Experimental): Since dose of RDEA3170 6 mg administered in fed or fasted state on Day 1 and Day 8.
  Interventions: Drug: RDEA3170 6 mg

INTERVENTIONS:
Drug: RDEA3170 4.5 mg
  Arms: Single Dose
Drug: RDEA3170 6 mg
  Arms: Single Dose; Single Dose Food Effect
Drug: RDEA3170 12 mg
  Arms: Multiple Dose; Single Dose

SUMMARY:
The purpose of this study is to examine the pharmacokinetic and pharmacodynamic effect of RDEA3170 when given as single or multiple doses

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body weight ≥ 50 kg (110 lbs.) and a body mass index ≥ 18 and ≤ 40 kg/m2.
* Subject has a Screening serum urate level 4 to 7 mg/dL
* Subject is free of any clinically significant disease or medical condition, per the Investigator's judgment.

Exclusion Criteria:

* Subject has a history or suspicion of kidney stones.
* Subject has undergone major surgery within 3 months prior to Screening.
* Subject donated blood or experienced significant blood loss within 12 weeks prior to Day 1 or gave a plasma donation within 4 weeks prior to Day 1.
* Subject has clinically unacceptable physical examination, per the Investigator's judgment.
* Subject has clinically relevant abnormalities in blood pressure, heart rate, or body temperature, per the Investigator's judgment.
* Subject has Screening clinical safety laboratory parameters (serum chemistry [other than serum creatinine and serum urate], hematology, coagulation or urinalysis) that are outside the normal limits and are considered clinically significant by the Investigator.
* Subject has a serum creatinine value above the upper limit of normal at the Screening visit.
* Subject has clinically relevant abnormalities in 12-lead electrocardiogram, per the Investigator's judgment.
* Subject has a history of cardiac abnormalities
* Subject has received any strong or moderate enzyme-inducing drug or product within 2 months prior to Day 1.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Days -1, 1, 5 and 9
  Single-dose Pharmacokinetic (PK) profile of RDEA3170 4.5 mg, 6 mg and 12 mg
Cmax | Days -1, 1 and 7
  Multiple-dose Pharmacokinetic (PK) profile of RDEA3170 12 mg
Cmax | Days -1, 1, 7 and 8
  Single-dose Pharmacokinetic (PK) profile of RDEA3170 6 mg under fed and fasted conditions
Time of Occurrence of maximum observed concentration (Tmax) | Days -1, 1, 5 and 9
  Single-dose Pharmacokinetic (PK) profile of RDEA3170 4.5 mg, 6 mg and 12 mg
Area under the plasma concentration time curve (AUC) | Days -1, 1, 5 and 9
  Single-dose Pharmacokinetic (PK) profile of RDEA3170 4.5 mg, 6 mg and 12 mg
Tmax | Days -1, 1 and 7
  Multiple-dose Pharmacokinetic (PK) profile of RDEA3170 12 mg
AUC | Days -1, 1 and 7
  Multiple-dose Pharmacokinetic (PK) profile of RDEA3170 12 mg
Tmax | Days -1, 1, 7 and 8
  Single-dose Pharmacokinetic (PK) profile of RDEA3170 6 mg under fed and fasted conditions
AUC | Days -1, 1, 7 and 8
  Single-dose Pharmacokinetic (PK) profile of RDEA3170 6 mg under fed and fasted conditions
Serum urate concentration | Days -1, 1, 5 and 9
  Single-dose Pharmacodynamic (PD) profile of RDEA3170 4.5 mg, 6 mg and 12 mg
Urine uric acid excretion amount | Days -1, 1, 5 and 9
  Single-dose Pharmacodynamic (PD) profile of RDEA3170 4.5 mg, 6 mg and 12 mg
Renal clearance of uric acid | Days -1, 1, 5 and 9
  Single-dose Pharmacodynamic (PD) profile of RDEA3170 4.5 mg, 6 mg and 12 mg
Fractional excretion of uric acid | Days -1, 1, 5 and 9
  Single-dose Pharmacodynamic (PD) profile of RDEA3170 4.5 mg, 6 mg and 12 mg
Serum urate concentration | Days -1, 1 and 7
  Multiple-dose Pharmacodynamic (PD) profile of RDEA3170 12 mg
Urine uric acid excretion amount | Days -1, 1 and 7
  Multiple-dose Pharmacodynamic (PD) profile of RDEA3170 12 mg
Renal clearance of uric acid | Days -1, 1 and 7
  Multiple-dose Pharmacodynamic (PD) profile of RDEA3170 12 mg
Fractional excretion of uric acid | Days -1, 1 and 7
  Multiple-dose Pharmacodynamic (PD) profile of RDEA3170 12 mg
Serum urate concentration | Days -1, 1, 7 and 8
  Single-dose Pharmacodynamic (PD) profile of RDEA3170 6 mg under fed and fasted conditions
Urine uric acid excretion amount | Days -1, 1, 7 and 8
  Single-dose Pharmacodynamic (PD) profile of RDEA3170 6 mg under fed and fasted conditions
Renal Clearance of Uric Acid | Days -1, 1, 7 and 8
  Single-dose Pharmacodynamic (PD) profile of RDEA3170 6 mg under fed and fasted conditions
Fractional excretion of uric acid | Days -1, 1, 7 and 8
  Single-dose Pharmacodynamic (PD) profile of RDEA3170 6 mg under fed and fasted conditions

SECONDARY OUTCOMES:
Incidence of Adverse Events in terms of changes in laboratory parameters | 6 weeks
Incidence of Adverse Events in terms of electrocardiogram parameters | 6 weeks
Incidence of Adverse Events in terms of vital signs | 6 weeks
Incidence of Adverse Events in terms of physical examination findings | 6 weeks
Apparent terminal half-life (t1/2) | Days -1, 1, 5 and 9
  Single-dose Pharmacokinetic (PK) profile of RDEA3170 4.5 mg, 6 mg and 12 mg from plasma and urine
t1/2 | Days -1, 1, 7 and 8
  Single-dose Pharmacokinetic (PK) profile of RDEA3170 6 mg under fed and fasted conditions
t1/2 | Days -1, 1 and 7
  Multiple-dose Pharmacokinetic (PK) profile of RDEA3170 12 mg from plasma and urine

CONTACTS AND LOCATIONS:
Overall Officials: J. Hall, MD, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Austin, Texas, United States